CLINICAL TRIAL: NCT05014802
Title: Baseline Atrial Fibrosis Predicts Risk for Post-operative Atrial Fibrillation in Patients Undergoing Cardiac Surgery: A Pilot Study for SAPPORO-AF
Brief Title: Baseline Atrial Fibrosis Predicts Risk for Post-operative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-622
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation; Atrial Arrhythmia; Atrial Flutter; Atrial Tachycardia
Keywords: Atrial Fibrosis; Cardiac Magnetic Resonance Imaging; Cardiac surgery
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate and compare the incidence of atrial arrhythmias (including Post-Operative Atrial Fibrillation (POAF), atrial flutter, and atrial tachycardia) stratified by baseline Utah fibrosis stages and overall fibrosis (%) of the left atrial wall area. The investigators hypothesize that patients with a higher baseline Utah fibrosis staging will experience a higher incidence of POAF.

The study also aims to evaluate and compare the in-hospital mortality, length-of-stay (LOS), complication rates (strokes, pneumonia, respiratory failure etc.) of the different Utah fibrosis stage cohorts. Perform cost analysis and compare between patients with POAF and patients without POAF. The investigators hypothesize that patients experiencing POAF will have a higher mortality rate, longer LOS, greater complications, and therefore, additional hospital costs.

DETAILED DESCRIPTION:
The study is a a prospective, observational cohort study. 50 patients undergoing cardiac surgery (Coronary Artery Bypass Graft (CABG), valvular etc.) without a history of atrial fibrillation will be given a baseline Magnetic Resonance Imaging (MRI) upon which patients will be assigned Utah stages I-IV based on their left atrial fibrosis pattern. Overall fibrosis (%) of the left atrial wall area will also be collected. Patients will then undergo their planned surgeries receiving management adherent to current guidelines and standard of care procedures. Atrial arrhythmia incidence after surgical procedure will be collected using in-hospital telemetry or serial Electrocardiogram (ECG) from all patients in their respective cohorts. Cardiac surgery type, duration and any intraoperative complications will be recorded. Other clinical and relevant demographical data will be collected at admission and throughout patients' hospital stay.

All cardiac surgeries will be performed by experienced surgeons at Tulane Medical Center, Washington University Medical Center Barnes Jewish Hospital, and University Medical Center New Orleans, adhering to all relevant standard-of-care guidelines. MRI imaging will be performed by experienced technicians and operators at Tulane Medical Center, Washington University Medical Center Barnes Jewish Hospital, and University Medical Center New Orleans. MRI Utah fibrosis staging will be performed and assessed by experienced operators at MARREK, Inc., by using the Corview processing software with de-identified images.

The investigators expect a total recruitment of 50 subjects over a period of 6 months from the Tulane Medical Center Cardiology and Cardiothoracic Surgery Clinics, Washington University Medical Center Barnes Jewish Hospital Cardiology and Cardiothoracic Surgery Clinics, as well as University Medical Center New Orleans Cardiology and Cardiothoracic Surgery Clinics in order to complete the study. They expect to recruit 40 patients from Washington University Medical Center and 10 patients from either Tulane Medical Center or University Medical Center New Orleans.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 40 years of age or older
* Patients with no history of atrial arrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia) scheduled to undergo cardiac surgery (These surgeries include but are not limited to coronary artery bypass graft (CABG), valvular repair/reconstruction, aneurysm repair, and insertion of pacemaker).

Exclusion Criteria:

* Patients with a history of atrial arrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia)
* Patients with a history of cardiac or open chest surgery
* Patients with a history of catheter ablation
* Patients under the age of 40
* Patients with left ventricular assist device (LVAD) or scheduled to have LVAD implanted
* Patients who have previously undergone extracorporeal membrane oxygenation (ECMO)
* Patients who have undergone or will undergo heart transplantation
* Patients with any health related Late Gadolinium Enhancement (LGE)-MRI contraindications (including previous allergic reaction to gadolinium, pacemakers, defibrillators, other devices/implants contraindicated for MRI)
* Acute or chronic severe renal disease with a low glomerular filtration rate (GFR), <30 mL per minute per 1.73 m2 will be excluded from the trial. (A creatinine measurement should be available within the last 6 months. If not, a creatinine blood test will be drawn to assess for renal function before the MRI acquisition).
* Patients weighing > 300 lbs. (MRI image quality decreases due to increased body mass index)
* Patients currently pregnant or breastfeeding, or plan to become pregnant during the study period
* Patients with cognitive impairment preventing them from giving informed consent will be excluded from the study
* Patients who cannot read, speak, and/or understand English

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is any patient with no history of atrial arrhythmia scheduled to undergo cardiac surgery and meets other inclusion/exclusion criteria).
  Each Site:
  * Approximately 10 Patients from either Tulane Medical Center and/or University Medical Center New Orleans.
  * Approximately 40 Patients from Washington University Medical Center (Barnes Jewish Hospital).
  The PIs and co-PI will have access to recruit patients through their cardiology and cardiothoracic surgery clinics.
  Participants may also be recruited from the community by direct advertising; emails, TV, flyers posted in public places, as well as online postings to study-site affiliated websites, social media platforms (Facebook, Twitter, Instagram) and LinkedIn.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial arrhythmia in patients after cardiac surgery | 2 weeks
  The incidence of any atrial arrhythmia (atrial fibrillation, atrial flutter, atrial tachycardia etc.) from after their surgical procedure to their discharge from the hospital.
  Atrial arrhythmia is defined as any abnormal atrial rhythm episode continuing for more than 30 seconds, starting immediately after the patient arrives at the post-operation ICU. All atrial arrhythmia starting after the operation will be monitored and recorded. This will be measured using continuous telemetry and/or serial ECG monitoring.

SECONDARY OUTCOMES:
Rate of in-hospital mortality | 2 weeks
  In-hospital mortality is defined as patient death during any point of hospital stay following cardiac surgery. This will be measured through patients medical chart review.
Hospital and Intensive Care Unit (ICU) length of stay (LOS) | 2 weeks
  LOS is defined as duration from admission to discharge in days in the hospital and ICU. This will be measured through patients medical chart review.
Incidence of stroke | 2 weeks
  Stroke is defined as sudden loss of brain function caused by an interruption of blood supply to the brain either through an ischemic or hemorrhagic modality. This will be measured through patients medical chart review.
Incidence of acute respiratory failure | 2 weeks
  Acute respiratory failure is any decrease in respiratory function resulting in hypoxemia (low arterial oxygen levels), hypercapnia (elevated levels of carbon dioxide gas) or a combination of the two. This will be measured through patients medical chart review.
Incidence of sudden cardiac arrest | 2 weeks
  Sudden cardiac arrest is the abrupt loss of heart function, breathing and consciousness. This will be measured through patients medical chart review.
Incidence of shock | 2 weeks
  Shock is a critical condition brought on by the sudden drop in blood flow through the body. This will be measured through patients medical chart review.
Incidence of systemic or pulmonary embolism | 2 weeks
  An embolus is a blood clot that forms in the systemic or pulmonary circulation that jeopardizes normal blood flow to the area causing organ dysfunction. This will be measured through patients medical chart review.
Incidence of infection post surgery | 2 weeks
  Infection is the invasion and multiplication of microorganisms in any area of the body, specifically the heart, lungs, blood and gastrointestinal and urinary tract. This will be measured through patients medical chart review.
Hospitalization costs to the patient | 2 weeks
  All costs related to the current episode of hospitalization including procedures, medication, personnel and machine time, calculated prior to insurance or Medicaid/Medicare discount. This will be obtained through hospital billing department.

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Marrouche, MD, Principal Investigator — Tulane University
Locations (3):
- United States (3):
  - Tulane University Medical Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Washington University Barnes-Jewish Hospital, St Louis, Missouri